CLINICAL TRIAL: NCT04268147
Title: APDM Instrumented Data Exchange for Ataxia (IDEA) Study
Brief Title: Instrumented Data Exchange for Ataxia Study
Acronym: IDEA
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Pfizer (Industry); Biogen (Industry); APDM Wearable Technologies (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB18-1580
Record Dates: First submitted 2020-02-04; First posted 2020-02-13 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-05

CONDITIONS: Spinocerebellar Ataxia Type 1; Spinocerebellar Ataxia Type 2; Spinocerebellar Ataxia Type 3; Spinocerebellar Ataxia Type 6; Friedreich Ataxia
MeSH Terms: conditions — Spinocerebellar Ataxias; Machado-Joseph Disease; Friedreich Ataxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Spinocerebellar Ataxia-1: individuals with a genetically confirmed diagnosis of SCA-1
- Spinocerebellar Ataxia-2: individuals with a genetically confirmed diagnosis of SCA-2
- Spinocerebellar Ataxia-3: individuals with a genetically confirmed diagnosis of SCA-3
- Spinocerebellar Ataxia-6: individuals with a genetically confirmed diagnosis of SCA-6
- Freidreich's Ataxia: individuals with a genetically confirmed diagnosis of FA
- FA Controls: Healthy, age-matched controls
- SCA Controls: Healthy, age-matched controls

SUMMARY:
This research study is testing body-worn sensors to measure movement during simple tests of coordination, in order to evaluate the progression and severity of ataxia.

ELIGIBILITY:
Inclusion Criteria:

* SCA 1, 2, 3, 6, and FA with mutations in the pathogenic range confirmed from genetic testing
* SCA: aged 18-75 years
* FA: aged 12-30, diagnosed between ages 5-25
* community dwelling
* physically/cognitively capable of consenting/assenting and complying with the protocol based on investigator's judgement
* able to walk independently 10 yards without an assistive device
* able to sit or stand unassisted for 30 seconds
* no other neurological or musculoskeletal disorder that could affect mobility
* no other history of head injury, vestibular function, stroke, or other disorders that could affect mobility
* willing and able to participate in a 2-year study
* consent to be video recorded while performing study assessments

Exclusion Criteria:

* dementia that limits subjects' ability to follow directions
* pain that limits mobility
* SCA: enrolled in a clinical drug trial

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ataxia clinics
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
iSARA | 2 years
  measurements collected by wearable inertial sensors during instrumented Scale for the Assessment and Rating of Ataxia (iSARA)
SARA | 2 years
  Scale for the Assessment and Rating of Ataxia (SARA) measurements evaluated by clinician to measure severity of spinocerebellar ataxia through coordination, speech, stance, and gait
mFARS | 2 years
  modified Friedreich's Ataxia Rating Scale (mFARS) measurements evaluated by clinician compared to measure severity of Friedreich's ataxia through coordination, speech, stance, and gait
Daily Life (UChicago site ONLY) | 2 weeks
  APDM SmartSox technology used to measure daily life activity(movement, falls, etc.) of all University of Chicago subjects
Ataxia App on Watch/iPhone | 2 years
  Bi-weekly assessments completed on Ataxia Application for Apple Watches and iPhones. Data collected includes active monitoring of speech, stance, coordination, gait and patient-reported symptoms.
Patient-Reported Questionnaires of Health | 2 years
  Activities, Balance, and Confidence (ABC) Questionnaire; EQ-5D-5L Health Questionnaire; Modified Fatigue Impact Scale (MFIS-5); Activities of Daily Living (ADLs)
Falls Questionnaire | 2 years
  Automatic email sent out to subjects inquiring about any falls and near falls they have experienced during the past month
Functional Staging | 2 years
  Clinician evaluates severity of ataxia symptoms.
Timed 25 Foot Walk | 2 years
  Subjects walk for 25 feet, as quickly and safely as possible, while being timed

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California-Los Angeles, Los Angeles, California
  - The University of Chicago, Chicago, Illinois
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Mass General Hospital, Boston, Massachusetts
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No